CLINICAL TRIAL: NCT00001698
Title: Randomized, Double Blind, Placebo-Controlled, Phase IIB Trial of Ketorolac Mouth Rinse Evaluating the Effect of Cyclooxygenase Inhibition on Oropharyngeal Leukoplakia: Collaborative Study of the NCI, NIDCD and the NIDCR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980118; 98-C-0118
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-06

CONDITIONS: Leukoplakia; Periodontal Disease
Keywords: Chemoprevention; Direct Epithelial Delivery; Tobacco-induced Cancer; Field Cancerization
MeSH Terms: conditions — Leukoplakia; Periodontal Diseases

INTERVENTIONS:
Drug: Ketorolac Rinse

SUMMARY:
In Phase II trials, treatment with ketorolac tromethamine oral rinse has been shown to block periodontal disease progression even in the absence of standard clinical intervention such as scaling and root planing which is routinely done to reduce the periodontal pathogen load that is driving the local destructive host inflammatory response. Resolution of periodontal disease has a favorable effect on normalizing the cellular and biochemical indices of inflammation as reflected by histological changes as well as the levels of prostaglandin E2 (PGE2) and interleukin I beta (IL-1beta). In this trial, we will prospectively evaluate if eliminating the inflammatory process (via inhibition of PGE2 biosynthesis) in the oral cavity has a favorable impact on reversing oropharyngeal leukoplakia. To test this hypothesis, up to 57 prospectively identified individuals with objective findings of oropharyngeal leukoplakia will be randomized to receive either a mouth rinse containing ketorolac or placebo. Ketorolac is a 7-fold selective inhibitor of cyclooxygenase-2 (Cox-2), which has been designed for local delivery to maximize the drug exposure to critical oral target tissues while minimizing gastric and systemic exposure to the drug. All responses will be determined at the three month completion of trial using the response criteria developed at MD Anderson Cancer Center. The drug will be given for three months and then all the patients will be followed for one additional month off all oral treatment to observe for late side effects. Based on the analysis of oral exam and photographically documented change in the pretreatment area of leukoplakia, the response of all patients will be determined.

The evaluation of the outcome will include a measurable secondary endpoint consisting of an assessment of histological change as determined by serial punch biopsies of the oral cavity. In addition, a panel of carcinogenesis and inflammatory markers will be serially measured at baseline, at one month follow up or at study conclusion. In the residual tissue, other bioassays will be evaluated to determine their suitability as intermediate endpoint markers. The purpose of this study is a preliminary evaluation of the effectiveness of ketorolac as a potential chemoprevention agent for oropharyngeal cancer. If ketorolac administration in this preliminary Phase IIB trial is associated with reversal of leukoplakia, then a definitive Phase III chemoprevention trial with a cancer reduction endpoint (most likely in a cooperative group-type setting) may be the next validation step.

DETAILED DESCRIPTION:
In Phase II trials, treatment with ketorolac tromethamine oral rinse has been shown to block periodontal disease progression even in the absence of standard clinical intervention such as scaling and root planing which is routinely done to reduce the periodontal pathogen load that is driving the local destructive host inflammatory response. Resolution of periodontal disease has a favorable effect on normalizing the cellular and biochemical indices of inflammation as reflected by histological changes as well as the levels of prostaglandin E2 (PGE2) and interleukin I beta (IL-1beta). In this trial, we will prospectively evaluate if eliminating the inflammatory process (via inhibition of PGE2 biosynthesis) in the oral cavity has a favorable impact on reversing oropharyngeal leukoplakia. To test this hypothesis, up to 57 prospectively identified individuals with objective findings of oropharyngeal leukoplakia will be randomized to receive either a mouth rinse containing ketorolac or placebo. Ketorolac is a 7-fold selective inhibitor of cyclooxygenase-2 (Cox-2), which has been designed for local delivery to maximize the drug exposure to critical oral target tissues while minimizing gastric and systemic exposure to the drug. All responses will be determined at the three month completion of trial using the response criteria developed at MD Anderson Cancer Center. The drug will be given for three months and then all the patients will be followed for one additional month off all oral treatment to observe for late side effects. Based on the analysis of oral exam and photographically documented change in the pretreatment area of leukoplakia, the response of all patients will be determined.

The evaluation of the outcome will include a measurable secondary endpoint consisting of an assessment of histological change as determined by serial punch biopsies of the oral cavity. In addition, a panel of carcinogenesis and inflammatory markers will be serially measured at baseline, at one month follow up or at study conclusion. In the residual tissue, other bioassays will be evaluated to determine their suitability as intermediate endpoint markers. The purpose of this study is a preliminary evaluation of the effectiveness of ketorolac as a potential chemoprevention agent for oropharyngeal cancer. If ketorolac administration in this preliminary Phase IIB trial is associated with reversal of leukoplakia, then a definitive Phase III chemoprevention trial with a cancer reduction endpoint (most likely in a cooperative group-type setting) may be the next validation step.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must have objective evidence of oral leukoplakia. This includes subjects who have had a previous diagnosis of head and neck or oral cancer, who are currently free of evidence of known cancer for at least three months.

Patients must have bidimensionally measurable lesions.

Patients must consent to serial photography and biopsy to document response to treatment.

All patients old enough to give their own informed consent (greater than or equal to 18 years old) are eligible.

Subjects must be excellent performance status (Performance Status 0-1).

In addition, they must be otherwise medically fit in the opinion of the PI with no other uncontrolled medical conditions.

EXCLUSION CRITERIA:

Patients with a hypersensitivity to aspirin, lidocaine or non-steroid anti-inflammatory agents or retinoids will be ineligible.

Patients using antibiotics, steroids, NSAID, aspirin, probenecid or antihistamines for an extended regimen of at least 10 or more consecutive days, or any immunosuppressants, anticoagulants, dilantin, lithium, methotrexate, phenothiazines, investigational drugs with pharmacological activity that could compromise the test product safety during the 30 days immediately preceding the first treatment visit.

Patients with serious or debilitating oral conditions that require extensive dental procedures in order to safely participate in this trial. This trial does not envision the need to do dental procedures (such as root canal or gingival procedure) in order to allow a potential participant to enroll on this study.

Individuals with a social or psychiatric situation interfering with study compliance or an unwillingness to undergo the serial oral biopsies will be excluded.

Patients with compromised respiratory function manifested by shortness of breath with mild exertion or dependency on supplemental oxygen.

Patients with compromised cardiovascular status including poorly controlled angina or congestive heart failure.

ELIGIBILITY FOR ORAL IMAGING SUBSTUDY:

Participation in this substudy requires that patients be enrolled in the parent trial.

Subjects must have given their consent and signed supplemental informed consent for the pilot study involving oral imaging.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57
Dates: Start 1998-06; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute (NCI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Cavanaugh PF Jr, Meredith MP, Buchanan W, Doyle MJ, Reddy MS, Jeffcoat MK. Coordinate production of PGE2 and IL-1 beta in the gingival crevicular fluid of adults with periodontitis: its relationship to alveolar bone loss and disruption by twice daily treatment with ketorolac tromethamine oral rinse. J Periodontal Res. 1998 Feb;33(2):75-82. doi: 10.1111/j.1600-0765.1998.tb02295.x. PMID 9553866
- [Background] Hong WK, Sporn MB. Recent advances in chemoprevention of cancer. Science. 1997 Nov 7;278(5340):1073-7. doi: 10.1126/science.278.5340.1073. PMID 9353183
- [Background] Potter M. Experimental plasmacytomagenesis in mice. Hematol Oncol Clin North Am. 1997 Apr;11(2):323-47. doi: 10.1016/s0889-8588(05)70434-2. PMID 9137973